CLINICAL TRIAL: NCT02722122
Title: A Proof-of-Concept, Open Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Exploratory Efficacy Parameters of AIR DNase™in Patients With Cystic Fibrosis Previously Treated With Pulmozyme®
Brief Title: Study to Evaluate the Safety,Tolerability, Pharmacokinetics and Exploratory Efficacy Parameters of AIR DNase™in Patients With Cystic Fibrosis Previously Treated With Pulmozyme®
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Protalix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PB-110-CF02
Record Dates: First submitted 2016-03-23; First posted 2016-03-29 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; CF; AIR DNase™; Digestive System Diseases; Genetic Diseases, Inborn; Infant, New born, Diseases; Lung diseases; Pancreatic Diseases; Respiratory Tract Diseases
MeSH Terms: conditions — Cystic Fibrosis; Digestive System Diseases; Genetic Diseases, Inborn; Disease; Lung Diseases; Pancreatic Diseases; Respiratory Tract Diseases

ARMS (1):
- AIR DNase™ 2.5 mg (Experimental): 2.5 mg of AIR DNase™ administered once daily via inhalation for 28 days
  Interventions: Drug: AIR DNase™

INTERVENTIONS:
Drug: AIR DNase™

SUMMARY:
This study evaluates the Safety,Tolerability, Pharmacokinetics and Exploratory Efficacy Parameters of AIR DNase™in Patients with Cystic Fibrosis previously treated with Pulmozyme®.

DETAILED DESCRIPTION:
This is a proof-of-concept, open label study, to evaluate the safety, tolerability, pharmacokinetics and exploratory efficacy of 2.5 mg AIR DNase TM administered once daily for 28 days via inhalation to Cystic Fibrosis subjects who have previously been treated with Pulmozyme®.

This multicenter study will be conducted in approximately 10 sites and will enroll up to 15 subjects.

ELIGIBILITY:
Main Inclusion Criteria:

1. Age ≥ 12 years of age (inclusive) at the time of screening
2. Weight ≥ 36 kg
3. Prior confirmed diagnosis of CF
4. At least 4 months treatment with Pulmozyme® prior to screening.
5. The subject is medically stable for at least one month prior to the screening visit.
6. Stable inhaled regimen of either: antibiotics, steroids, hypertonic saline at least four months prior to screening visit.
7. FEV1 of >40% and <90% and FVC ≥ 40% of predicted normal for age, gender, and height at screening .
8. Female and male subjects whose co-partners are of child bearing potential must agree to use two medically acceptable methods of contraception, not including the rhythm method.
9. Be willing and able to adhere to the study visit schedule and other protocol requirements
10. Be willing and able to provide voluntary written informed consent

Main Exclusion Criteria:

1. Has a history of lung transplantation.
2. Female subjects who are pregnant or lactating.
3. History of severe or unexplained adverse reactions during aerosol delivery of any medicinal product.
4. History or presence of hypersensitivity or reaction to inhaled proteins.
5. Participation in another clinical trial within 60 days prior to screening.
6. Presence of any medical, emotional, behavioral or psychological condition that in the judgment of the Investigator would interfere with the subject's safety or compliance with the requirements of the study.
7. Have positive serology for human immunodeficiency virus (HIV) or Hepatitis B or Hepatitis C infection.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Adverse events following daily administration of AIR DNase™ | 56 days
  Adverse events from subject reporting or other assessments

SECONDARY OUTCOMES:
Area under the curve | Up to 4 hours
  AIR DNase concentrations measured at 0, 0.25, 0.5, 0.75, 1, 1.5, 2, and 4 hours
Change from baseline to end of AIR DNase™ treatment in FEV1 | Baseline and 28 days
Change from baseline to end of AIR DNase™ treatment in FVC | Baseline and 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Einat Dekel, DVM, Study Director — Sr. Director Clinical Development
Locations (5):
- Israel (5):
  - Carmel MC, Haifa
  - Rambam MC, Haifa
  - Hadassah MC, Jerusalem
  - Schneider MC, Petah Tikva
  - Sheba MC, Ramat Gan